CLINICAL TRIAL: NCT03678831
Title: Characterization of Bone Marrow Adipocytes in Osteoarthritic and Post-menopausal Patients: a Comparative Study With Adipocytes From Subcutaneous Adipose Tissue
Brief Title: Characteristics of Marrow Fatty Cells in the Ageing of Bone and Joints, Osteoarthritis and Osteoporosis
Acronym: MEDADIPO
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: MSDAVENIR Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017_59; 2018-A00660-55 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Knee; Prosthesis User
Keywords: Osteoarthritis; prosthetic surgery of the knee; obesity; type 2 diabetes; bone marrow fat
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Obesity; Diabetes Mellitus, Type 2 | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arthritic patients with knee prosthetic replace: Arthritic post-menopausal patients with knee prosthetic replacement Each patient is her own control since the two cell types are compared within the same patient The main criteria is based on a comparison of two cell types from the same patient. The secondary criteria are based on a comparison of cell types according to a grouping of patients according to different metabolic parameters.
  Interventions: Procedure: tissue

INTERVENTIONS:
Procedure: tissue — Adipocyte isolation from distal femoral epiphysis and subcutaneous adipose tissue at the surgery site; classical piece removal during prosthetic replacement of the knee

SUMMARY:
Obesity and other associated complications promote the development and the progression of osteoarthritis. The subcutaneous and abdominal fat release several factors that alter bone and the cartilage. The role of the marrow fat in close connection with bone has not been defined yet, whereas cellular and animal models indicate that this fat depot modifies bone and cartilage.

The aim of the study is to define if the marrow fat produces more joint-altering factors by comparison with subcutaneous fat. This fat depot can be characterized from removed pieces during the prosthetic surgery of the knee. Measuring before surgery the body weight, waist and hip circumferences, blood pressure, glucose, insulin and lipids in blood will also allow to determine if obesity and/or type 2 diabetes make this fat more dangerous for the joint. Such research will allow the elaboration of new therapeutic strategies in osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal woman
* with a symptomatic knee osteoarthritis requiring prosthesis
* able to handle general anaesthesia
* having given her consent
* able to understand the constraints associated with the study
* with health insurance
* able to understand the French language

Exclusion Criteria:

* with refusal to participate to the study
* more than 85-year-old
* with bone pathologies other than osteoarthritis or osteoporosis
* with active infection
* with evolving cancer
* with haematopoietic pathologies such as haemoglobin pathologies
* with thyroid pathologies
* with type 1 diabetes
* with anti-osteoporotic treatments (bisphosphonates, strontium ranelate, teriparatide, denosumab) except calcium and vitamin D supplementation or hormone replacement.
* with replacement of prosthesis
* with previous surgery at the surgery site

  --with a current participation to another study
* with guardianship
* with deprived liberty

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Arthritic post-menopausal patients with knee prosthetic replacement
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Expression levels in femoral spinal adipocytes of mRNAs of 18 genes compared to those of adipocytes isolated from the subcutaneous adipose tissue in the same patient | at 3 months

SECONDARY OUTCOMES:
the intra patients difference of the expression level of medullary adipocytes mRNA compared to that of subcutaneous adipocytes according to Obesity state (normal vs overweight vs obese) as defined using BMI | at 3 months
the intra patients difference of the expression level of medullary adipocytes mRNA compared to that of subcutaneous adipocytes according to Central obesity (yes or no) as defined using the waist-to-hip ratio | at 3 months
the intra patients difference of the expression level of medullary adipocytes mRNA compared to that of subcutaneous adipocytes according to Presence or absence of systemic insulin-resistance as measured using the HOMA-IR index | at 3 months
  the Homeostatic Model Assessment of Insulin Resistance(HOMA-IR index)Healthy Range: 1.0 (0.5-1.4) Less than 1.0 means you are insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance. Above 2.9 indicates significant insulin resistance.
the intra patients difference of the expression level of medullary adipocytes mRNA compared to that of subcutaneous adipocytesaccording to Presence or absence of chronic uncontrolled hyperglycaemia as measured using HbA1c plasma levels | at 3 months
the intra patients difference of the expression level of medullary adipocytes mRNA compared to that of subcutaneous adipocytes according to presence or absence of metabolic syndrome | at 3 months
  metabolic syndrome as defined by the presence of at least three of the following criteria: large waist circumference, decrease in HDL-cholesterol, hypertriglyceridemia, elevated fasting glycaemia, elevated blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Pasquier, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France